CLINICAL TRIAL: NCT04546646
Title: Effects of Elastic Band Exercises on Physical Performance in Community Dwelling Elderly With Locomotive Syndrome
Brief Title: Elastic Band Exercises and Locomotive Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/20/1044 Sania Anwaar
Record Dates: First submitted 2020-09-04; First posted 2020-09-14 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Locomotive Syndrome
Keywords: Locomotive Syndrome; Geriatric; Elastic Band Resistance Exercises.

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A (Elastic Band Exercises) (Experimental): Warm up: for 10 min, Exercise: Lower limb exercises using elastic band for 30 min. Cool down: Self-stretches 5 min.
  Interventions: Other: Elastic Band Exercises
- GROUP - B (No Intervention) (No Intervention): Routine activities of daily living

INTERVENTIONS:
Other: Elastic Band Exercises — Resistance exercise will be performed using theraband. The color of the band denotes the degree of elasticity and resistance level(yellow , red ,green ,blue, black or silver).Exercise load in terms of individual yielding elasticity (band color) in resistance training will set at a level that a patient perceived as somewhat hard, which is equivalent to a 13-grade rating (moderate intensity exercise) on the RPE, According to American College of Sports Medicine. For each exercise movement 3 sets of 10 repetitions of gentle concentric and eccentric contractions through the full range of motion will be slowly performed using a yellow Thera band initially. The exercise intensity will be increased when the patient is able to achieve a perceived yield strength corresponding to a 13- grade rating on the RPE scale.
  Arms: GROUP A (Elastic Band Exercises)

SUMMARY:
Locomotive syndrome is described as a condition in which mobility functions such as gait or Sit-to-stand are decreased due to impairment of the locomotive organs. Progression of locomotion syndrome causes limitation in carrying out activities of daily living (ADL) independently. So interventions are required to limit the progression of the syndrome and to sustain the functions of locomotive organs. This study will be a randomized controlled trial in which elastic band exercises are used to enhance the physical performance of community-dwelling elderly with locomotive syndrome and changes will be recorded using different methods and tools. Non-probability convenient sampling technique will be used to collect the data. The sample size of 24 patients will be taken in this study. Patients will be randomly allocated into two different groups through sealed envelope method. Group A will be treated with elastic band exercises and Group B will have no intervention. Short physical performance battery protocol and score sheet tool will be used as outcome measure tool. Participants of both groups will be pre-tested before the application of interventional techniques and post-tested after the application of respective interventions after 3 months. Data will be analyzed on SPSS 21.

DETAILED DESCRIPTION:
Locomotive syndrome is described as a condition in which mobility functions such as gait or Sit-to-stand are decreased due to impairment of the locomotive organs. Progression of locomotion syndrome causes limitation in carrying out activities of daily living (ADL) independently. So interventions are required to limit the progression of the syndrome and to sustain the functions of locomotive organs. Locomotive system of the body consist of 3 components which are Bones (support), joint and intervertebral discs(mobility, impact absorption) and muscular and nervous system (drive , control). Any dysfunction in these locomotive organs can lead to the development of pain, limited range of motion at joints muscle weakness and balance deficits. Common diseases of the locomotive organs which are non-traumatic etiology are chronic diseases disc degeneration, lower extremity cartilage degeneration and traumatic causes includes fractures due to osteoporosis.

Population of Japan is aging so rapidly 8-10% of people are 65 or above, and is already be seen as super aged society, it has great impact on social system including public health. Japanese did great work in this perspective and also the world .First described the term locomotive syndrome . Japanese Orthopedic Association (JOA) proposed the term of locomotive syndrome (LS) in 2007 to describe the conditions of patients with high-risk musculoskeletal diseases requiring Nursing care.GLFS-25 is geriatric locomotive function scale a screening tool developed by the JOA in 2012. A score >16 indicates the presence of locomotive syndrome. GFLS is used to Assess a participant's physical condition and lifestyle over a prior month. It is self-administered and comprehensive questionnaire having 25 items, which include questions related to pain, Activities of daily living (ADL),social function and mental health status. 25 points are Graded from 0 points(no impairment)to 4 points (severe impairment. The (SPPB )Short Physical Performance Battery Protocol And Score Sheet is commonly used To measure balance ,gait speed and lower limb strength and endurance. There is more rapid functional decline in lower extremities than in lower extremities in individuals with locomotive syndrome. SPPB score of 6 is a low performance score. Different types of intervention strategies are used for the strengthening of muscles in adults but as far as elderly individuals are concerned there is a need for the intervention which is effective, inexpensive ,easy and most importantly safe to execute. To strengthen the weakened musculature resistance exercises are commonly performed. Elastic bands are the bands or tubes of plastic material which can provide load or resistance in all directions. Elastic bands of different resistance. are available and their coloring shows strength levels. Force that an elastic band generate is directly proportional to its length. By changing the length and thickness of these bands their resistance levels can be increased or decreased. Depending on the brand of resistance band most common colors are yellow, green, red, blue, black, silver and gold with yellow being the lightest and gold the strongest. It is easy to adjust the resistance of elastic band in muscle strengthening so these are commonly used for rehabilitation treatment of disorders and sports injuries because of their low cost and simplicity. In addition to increase in physical performance elastic band exercises also decreases the depression and anxiety. It is difficult for the elderly population to adhere with a continued training so elastic band exercises can be incorporated in training which are easy and simple to perform. Almost all the exercises with elastic bands can be performed at any place while walking ,travelling and everywhere because no tool or equipment is required. Previous studies did not used elastic band exercises in community-dwelling elderly to increase the physical performance.

ELIGIBILITY:
Inclusion Criteria:

1. Age >60 years
2. Both genders
3. Greater than 16 score on Geriatric Locomotive Function Scale (GLFS)
4. Complaints related to legs and spine without disability in walking or going out.
5. Score of less than 45 in Berg Balance Scale.
6. Some difficulty in walking due to locomotive organ dysfunction.
7. Good communication and ability to perform activities of Short physical performance battery protocol.

Exclusion Criteria:

1. Persons with severe co-morbid conditins
2. Stroke
3. Cardiac failure
4. Cognitive impairment
5. Alzheimer's disease

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery Protocol and Score Sheet | 12 Weeks
  It is a clinician-rated physical measures that evaluates physical function in older adults. This assessment consist of 3 sub-scales: standing balance, gait , rising from chair . The assessment is scored on a 0-12 scale,with higher scores indicating better function. The SPPB does not require specific training ,is free to use and requires only a stopwatch and chair .

CONTACTS AND LOCATIONS:
Overall Officials: Danish Hassan, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akahane M, Yoshihara S, Maeyashiki A, Tanaka Y, Imamura T. Lifestyle factors are significantly associated with the locomotive syndrome: a cross-sectional study. BMC Geriatr. 2017 Oct 18;17(1):241. doi: 10.1186/s12877-017-0630-1. PMID 29047351
- [Background] Akai M, Doi T, Seichi A, Okuma Y, Ogata T, Iwaya T. Locomotive Syndrome: Operational Definition Based on a Questionnaire, and Exercise Interventions on Mobility Dysfunction in Elderly People. Clin Rev Bone Miner Metab. 2016;14:119-130. doi: 10.1007/s12018-016-9210-8. Epub 2016 Jun 3. PMID 27375372
- [Background] Iwaya T, Doi T, Seichi A, Hoshino Y, Ogata T, Akai M. Characteristics of disability in activity of daily living in elderly people associated with locomotive disorders. BMC Geriatr. 2017 Jul 26;17(1):165. doi: 10.1186/s12877-017-0543-z. PMID 28747158
- [Background] Kataoka H, Miyatake N, Ichikawa H, Arakawa Y, Mori Y. Relationship of locomotive syndrome with health-related quality of life among patients with obstructive sleep apnea syndrome. J Phys Ther Sci. 2017 Jul;29(7):1129-1133. doi: 10.1589/jpts.29.1129. Epub 2017 Jul 15. PMID 28744031
- [Background] Matsumoto H, Hagino H, Wada T, Kobayashi E. Locomotive syndrome presents a risk for falls and fractures in the elderly Japanese population. Osteoporos Sarcopenia. 2016 Sep;2(3):156-163. doi: 10.1016/j.afos.2016.06.001. Epub 2016 Jul 1. PMID 30775481